CLINICAL TRIAL: NCT03540719
Title: Surgical Management of Posterior Tibial Plateau Fractures
Acronym: Proxtib
Status: Completed | Type: Observational
Sponsor: Harm Hoekstra, prof. dr. (Other)
Responsible Party: Sponsor-Investigator, Harm Hoekstra, prof. dr., Prof. Dr. Harm Hoekstra, Universitaire Ziekenhuizen KU Leuven
Organization: Universitaire Ziekenhuizen KU Leuven (Other)
Other Study IDs: S60860
Record Dates: First submitted 2018-05-02; First posted 2018-05-30 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Tibial Fractures
Keywords: classification; questionnaires; open reduction; internal fixation
MeSH Terms: conditions — Tibial Fractures | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Osteosynthesis — Osteosynthesis of posterior tibial plateau fracture with a posterior tibial plateau plate

SUMMARY:
This protocol concerns an academic, multicentric, and prospective clinical trial. In this study the investigators will evaluate the recently approved WAVE-plate (7S Medical) for open reduction and internal fixation and buttressing of the posterior proximal tibial column via a posteromedial reversed L-shaped approach. The reversed L-shaped approach has been shown as a safe technique with adequate visualisation of the posterior tibial surface. The investigators will thoroughly evaluate all important clinical, radiological and functional variables. The functional outcome will be reported in patient reported outcome measures by means of the validated Knee injury and Osteoarthritis Outcome Score (KOOS).

ELIGIBILITY:
Inclusion Criteria:

* Tibial plateau fracture with involvement of posterior proximal tibial plateau (according to revised three-column classification), requiring osteosynthesis

Exclusion Criteria:

* Absent contact information
* living abroad and cannot participate in the follow-up visits
* non-functional leg prior to treatment/injury
* pathological fractures
* bilateral fractures

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient at emergency room and clinic of the department of traumatology.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Subjective evaluation: outcome | 1 year
  Total Knee injury and Osteoarthritis Outcome Score (KOOS) questionnaire to measure patient's opinion about his or her knee and the associatede problems.
Subjective evaluation: pain | 1 year
  Visual analogue scale (VAS) to indicate the daily pain level.
Clinical evaluation | 1 year
  Recording of demographic and fracture-related characteristics.
Radiographic evaluation | 1 year
  Parameters derived from CT and RX.

SECONDARY OUTCOMES:
Complications | 1-7 days post-operatively, 8 weeks, 12 weeks, 6 months, 9 months, 1 year
  Recording of complications: infection, nonunion, wound related problems, implant related complaints, compartment syndrome, neurological disorder, muscle atrophy and deep vein thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Harm Hoekstra, Prof. MD, Principal Investigator — UZ Leuven
Locations (4):
- Belgium (2):
  - UZ Brussel, Brussels
  - UZ Leuven, Leuven
- Erasmus MC Rotterdam, Rotterdam, Netherlands
- Luzerner Kantonsspital Luzern, Lucerne, Switzerland